CLINICAL TRIAL: NCT03775174
Title: Expanded Access to Mepsevii
Status: Available | Type: Expanded Access
Sponsor: Ultragenyx Pharmaceutical Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: UX003-EAP
Record Dates: First submitted 2018-12-11; First posted 2018-12-13 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: MPS VII; Mucopolysaccharidosis VII; Sly Syndrome
Keywords: Expanded Access; Compassionate Use
MeSH Terms: conditions — Mucopolysaccharidosis VII | interventions — vestronidase alfa

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Drug: Mepsevii
  Other Names: UX003; recombinant human beta-glucuronidase; rhGUS; vestronidase alfa

SUMMARY:
Individual patient expanded access requests may be considered for patients who have no other treatment options

DETAILED DESCRIPTION:
Expanded access may be available outside of the US in countries prior to approval by the local regulatory agencies. For full details, please visit the links provided below.

ELIGIBILITY:
Inclusion Criteria:

-

Exclusion Criteria:

-

Sex: All
Age Groups: Child, Adult, Older Adult

REFERENCES:
- See also: Access to Investigational Therapies / Requesting Access — https://www.ultragenyx.com/our-purpose/supporting-access-for-patients/?#investigational-therapies
- See also: Mepsevii Patient and Prescribing Information Page — https://www.mepsevii.com/en/